CLINICAL TRIAL: NCT04651855
Title: The Evaluation of the Effect of Wharton's Jelly Mesenchymal Stem Cells (WJMSCs) on the Immune System of Patients With Amyotrophic Lateral Sclerosis (ALS)
Brief Title: The Evaluation of the Effect of Mesenchymal Stem Cells on the Immune System of Patients With ALS
Acronym: ALSTEM
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Polski Bank Komorek Macierzystych JSC (PBKM) (Industry)
Collaborators: National Center for Research and Development, Poland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: ALSTEM
Record Dates: First submitted 2020-09-30; First posted 2020-12-03 (Actual); Last update posted 2022-05-03 (Actual); Status verified 2022-04

CONDITIONS: Amyotrophic Lateral Sclerosis
Keywords: Amyotrophic Lateral Sclerosis; Stem Cells
MeSH Terms: conditions — Amyotrophic Lateral Sclerosis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Treatment arm (Experimental): It is planned that IMP administration will be performed three times for each enrolled patient. IMP administration could be performed only if the patients does not have any contraindications for lumbar puncture.
  Interventions: Drug: Mesenchymal stem cells isolated from Wharton's jelly

INTERVENTIONS:
Drug: Mesenchymal stem cells isolated from Wharton's jelly — Intrathecal administration of mesenchymal stem cells

SUMMARY:
The objective of this study is to evaluate the safety of intrathecal administration of Wharton's Jelly Mesenchymal Stem Cells (WJMSC) and the impact on the immune system of patients with Amyotrophic Lateral Sclerosis.

DETAILED DESCRIPTION:
Clinical Phase: I/II

Population: Patients with Amyotrophic Lateral Sclerosis.

Project Design: One arm, non-blinded, open label study

Planned Sample Size: 20 patients

Investigational Medicinal Product: active IMP - mesenchymal stem cells isolated from Wharton's jelly

Screening:

Three visits on site to check the eligibility criteria (around 90, 60 and 30 days before first IMP administration)

Treatment (IMP administration):

Each patient will receive IMP three times: on baseline (day 0), 30 and 60 days after baseline (+/- 7 days).

Administration route: intrathecal

Follow up:

Duration: 18 months after first IMP administration Four on-site visits (3, 6, 9, 12 months after first IMP administration) and seven phone visits (4, 5, 7, 8, 10, 11 and 18 months after first IMP administration)

ELIGIBILITY:
Inclusion Criteria:

1. Adult patients (at least 18 years old)
2. The minimum patient's weight is not less than 40 kg
3. Diagnosis of sporadic ALS, definite or probable, as defined by El Escorial World Federation of Neurology criteria
4. History of ALS symptoms less than 2 years duration from the first symptoms of the disease
5. More than 6 months from diagnosis of the disease
6. Disease progression at 6 past months at least 3 points during this period of time assessed in ALSFRS-R scale
7. ALSFRS-R scale of at least 30 at screening appointment
8. Forced vital capacity >70% of predicted value for age, gender and height
9. Treatment with stable dose of riluzole(2x 50mg per 24h) before baseline visit (for at least 1 month)
10. Capable of providing written informed consent
11. Able to comply with study requirements and willing to follow all study procedures and follow-up visits
12. Women of child-bearing age and men with partners of child-bearing potential must agree to use two forms of contraceptive therapy throughout the course of the trial
13. Women of child-bearing age must undergo pregnancy test
14. Polish-language native speakers or patients who are proficient in the Polish language

Exclusion Criteria:

1. Pregnancy or breastfeeding
2. Tracheostomy
3. Ventilator dependence
4. Renal disease with creatinine >2mg/dl
5. Liver disease with ALT, AST or GGTP 2-fold higher than upper normal limit
6. Positive test for HBV, HCV, HIV with NAT method
7. Positive tests for syphilis
8. Any other clinically significant abnormalities on laboratory evaluation
9. Any condition that would compromise ability of undergoing lumbar puncture
10. Active systemic disease
11. Autoimmune disease (Hashimoto disease under control is allowed)
12. Uncontrolled diabetes (HbA1c > 8%)
13. Pulmonary disease that could affect interpretation of spirometry
14. Neurological concomitant disease
15. Unstable psychiatric concomitant disease
16. High risk of suicide
17. History of substance abuse within past year
18. History of malignancy, within the previous 5 years, including melanoma with exception of localized skin cancers
19. Any other clinically significant medical condition that can compromise patient's safety in the opinion of the investigator
20. Treatment with immunomodulatory drugs (for example immunoglobulins, corticosteroids or other immunosuppressant) in last 6 months
21. Participation in another clinical trial in last 6 months
22. Previous cellular therapy of any kind
23. Hypersensitivity to any component used in the cell culture
24. Nuchal rigidity and other signs of meningitis
25. Patients on chronic anticoagulation treatment (heparin/ warfarin/acenocoumarol/(N)OAC)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 20 (Actual)
Dates: Start 2020-12-02 (Actual); Primary Completion 2022-03-08 (Actual); Study Completion 2023-04 (Estimated)

PRIMARY OUTCOMES:
The number of (S)AESI [(Serious) Adverse Event of Special Interest] | 3 month FU (follow-up)
  (S)AESI are defined as:
  1. Meningitis and encephalitis.
  2. Toxic encephalopathy.
  3. High fever >39⁰C.
  4. Epileptic seizures that are not connected to conditions above (meningitis, encephalitis, toxic encephalopathy, high fever).

SECONDARY OUTCOMES:
Disease progression | screening, run-in period (-60 day and -30 day), at baseline and at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 and 18 month FU
  Disease progression assessed in ALSFRS-R scale (Revised Amyotrophic Lateral Sclerosis Functional Rating Scale). Higher scores mean a better outcome.
  Minimum: 0 points Maximum: 48 points
Pulmonary function decline | screening, run-in period (-60 day and -30 day), at baseline and at 1, 2, 3, 6, 9 and 12 month FU.
  Pulmonary function decline assessed in spirometry (forced vital capacity)
Muscle strength decline | screening, run-in period (-60 day and -30 day), at baseline and at 1, 2, 3, 6, 9 and 12 month FU
  Muscle strength decline
Upper motor neuron function | screening, run-in period (-60 day and -30 day), at baseline and at 1, 2, 3, 6, 9 and 12 month FU
  Upper motor neuron function assessed in UMNS scale (Upper Motor Neuron Scale). Best outcome 16 points, worst outcomes: 0 points and 48 points Minimum: 0 points Maximum: 48 points
Cognitive function | screening and 12 month FU
  Cognitive function assessed in ECAS (The Edinburgh Cognitive and Behavioural ALS Screen). Higher scores mean a better outcome.
  Minimum: 0 points Maximum: 136 points
Quality of life changes | screening, run-in period (-60 day and -30 day), at baseline and at 1, 2, 3, 4, 5, 6, 7, 8, 9, 10, 11, 12 and 18 month FU
  Quality of life changes, assessed by EQ-5D questionnaire - standardized instrument for measuring generic health status. Higher scores mean a better outcome.
The change of defined cytokines, chemokines, growth factors and pNFH (phosphorylated neurofilament heavy chain) level in CSF (Cerebrospinal fluid) | run-in visit (-60 day), at baseline and at 1, 2 and 6 month FU (12 month FU optional)
  The change of defined cytokines, chemokines, growth factors and pNFH level assessed in the samples of CSF
The change of defined cytokines, chemokines level in blood | screening visit, run-in period (-60 day and -30 day), at baseline and at 1, 2, 3, 6, 9 and 12 month FU.
  The change of defined cytokines, chemokines level assessed in the samples of blood serum
The change of creatinine and p75ECD level in urine | screening visit, run-in period (-60 day and -30 day), at baseline and at 1, 2, 3, 6, 9 and 12 month FU.
  The change of creatinine and p75ECD level
Muscle function changes | baseline and at 1, 2, 6 and 12 month FU
  Muscle function changes, assessed based on EMG examination (Electrophysiological examination of the muscle - MUNIX - motor unit number estimation)
The change of the brain visualization | run-in visit (-60 day), 6 and 12 month FU
  The change of the brain visualization in MRI (T1, T2 and DTI)
SAE (Serious Adverse Event)/AE (Adverse Event) and (S)AESI | 18 month FU
  The number of SAE/AE and (S)AESI - defined as in Outcome 1
Survival period to disease progression | 18 month FU
  The number of days from patients randomization to the end of the patients participation in the trial or to the one of the following:
  * PAV (permanent assisted ventilation)
  * Tracheostomy
  * Death
Mortality rate | 18 month FU
  Percentage of deaths in the entire study population.

CONTACTS AND LOCATIONS:
Locations (1):
- JST sp. z o.o., Częstochowa, Poland

IPD SHARING:
Plan to Share IPD: Undecided